CLINICAL TRIAL: NCT00218335
Title: A Network & Dyad HIV Prevention Intervention for IDU's
Brief Title: A Network & Dyad HIV Prevention Intervention for IDU's - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Carl Latkin, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DESPR DA016555-1; 5R01DA016555-05 (NIH); 5R01DA016555-04 (NIH); 5R01DA016555-03 (NIH); 3R01DA016555-03S1 (NIH); 3R01DA016555-02S1 (NIH); 5R01DA016555-02 (NIH); 3R01DA016555-01S1 (NIH); 1R01DA016555-01 (NIH); R01-16555-1; NIDA-16555-1; NCT00597155 (obsolete NCT alias)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-03

CONDITIONS: HIV; Hepatitis
Keywords: HIV prevention Intervention, injection drug user,peer-oriented, randomized controlled trial, social network
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Condition (Experimental): Participants were trained to be Health Educators. The intervention focused on HIV risk reduction by teaching knowledge and skills to reduce injection, drug splitting, and sex risk, and by teaching communication skills to conduct outreach to personal risk network members. The intervention consisted of five group-based sessions, one individual session, and one dyad session with a risk network member.
  Interventions: Behavioral: Intervention Condition
- Control Condition (Active Comparator): The control condition focused on injection drug-use related topics (e.g. HIV testing, Hepatitis C and drug overdose). The sessions were educational and did not include skills training. The control condition consisted of five group-based sessions.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Intervention Condition — In the intervention Condition participants were trained to be Health Educators. The intervention focused on HIV risk reduction by teaching knowledge and skills to reduce injection, drug splitting, and sex risk, and by teaching communication skills to conduct outreach to personal risk network members. The intervention consisted of five group-based sessions, one individual session, and one dyad session with a risk network member.
  Other Names: STEP into action
  Arms: Intervention Condition
Behavioral: Control Condition — The control condition focused on injection drug-use related topics (e.g. HIV testing, Hepatitis C and drug overdose). The sessions were educational and did not include skills training. The control condition consisted of five group-based sessions.
  Arms: Control Condition

SUMMARY:
The purpose of this study is to evaluate a peer-based HIV prevention intervention that targets active injection drug users and their drug and sex partners.

DETAILED DESCRIPTION:
HIV seroincidence among injection drug users remains high, with unprotected sexual contact substantially contributing to new HIV infections among injection drug users (IDUs). Interventions that are culturally competent and target drug users' main sex and drug partners may be especially effective for HIV/STI and HCV control and prevention.

The intervention to be tested in this study draws upon theoretical and empirical evidence suggesting that peer educator programs can have significant effects on the risk-related behaviors of both the educators and the peers whom they educate. Specifically, through group and individual focused sessions, participants learn and practice skills designed to reduce drug and sex related risk behaviors. Furthermore, individuals and their main risk partners attend a training session that focuses on risk reduction within their relationship.

ELIGIBILITY:
Inclusion Criteria:

(i)Self reported injection drug use within the prior 6 months; (ii)Willingness to invite a risk network member into the study and to talk about HIV prevention; (iii)Age 18 or older

Exclusion Criteria:

* Not concurrently enrolled in another HIV prevention intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2003-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Lighthouse, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from March 2004 to March 2006. Two types of participants were recruited: Index and Risk Network Members. Recruitment methods for Index included: street-based outreach, word of mouth, ads and referrals from community agencies. During the Index's baseline interview, a list of Risk Network Members was generated.
Pre-assignment Details: Two types of participants were enrolled in the study- index and networks. Networks did not go through the intervention or control condition. Index participants had to refer a network member AND show up for randomization in order to be enrolled in the intervention or control condition.
Groups:
- Intervention Condition: Index participants in the intervention condition were trained to be Health Educators. The intervention focused on HIV risk reduction by teaching knowledge and skills to reduce injection, drug splitting, and sex risk, and by teaching communication skills to conduct outreach to personal risk network members. The intervention consisted of five group-based sessions, one individual session, and one dyad session with a risk network member.
- Control Condition: Index participants in the control condition attended groups that focused on injection drug-use related topics (e.g. HIV testing, Hepatitis C and drug overdose). The sessions were educational and did not include skills training. The control condition consisted of five group-based sessions.
- Non-Randomized Baseline Index Participants: Those Index participants that completed a baseline interview but were not randomized into the intervention or control condition.
- Risk Network Members: Individuals from the personal social networks of the index participants who inject or are the sexual partners of the index participant
Period: Overall Study
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Started | 114 | 113 | 373 | 424
6 Month Follow-up | 103 | 99 | 219 | 301
12 Month Follow-up | 95 | 102 | 244 | 303
18 Month Follow-up | 101 | 108 | 296 | 368
Completed | 108 | 110 | 319 | 388
Not Completed | 6 | 3 | 54 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members | Total
Number analyzed (Participants) | 114 | 113 | 373 | 424 | 1024
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 114 | 113 | 372 | 422 | 1021
  >=65 years | 0 | 0 | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 43.9 (8) | 43.0 (7) | 42.4 (9) | 43.7 (8) | 43.2 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 130 | 170 | 403
  Male | 63 | 61 | 243 | 254 | 621
Region of Enrollment [Number; unit: participants]
  United States | 114 | 113 | 373 | 424 | 1024

OUTCOME MEASURES:

1. Primary Outcome: Any Sex Risk
Time Frame: 6 months
Population: The discrepancy between participant flow and number of participants analyzed is due to missing data and skip patterns employed during data collection.
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 101 | 98 | 217 | 298
participants | 48 | 62 | 119 | 179

2. Primary Outcome: Talked About HIV-related Topics With Drug Buddies (in the Past Month)
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 95 | 87 | 206 | 252
participants | 80 | 54 | 108 | 104

3. Primary Outcome: Showed a Needleless Syringe to Drug Buddies
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 103 | 99 | 219 | 300
participants | 85 | 18 | 32 | 49

4. Primary Outcome: Talked About Responding to Overdose to Drug Buddies
Time Frame: 6 months
Population: Data for this outcome was only measured among randomized participants (intervention and control participants), not among non-randomized and network participants. The discrepancy between participant flow and number of participants analyzed is due to missing data and skip patterns employed during data collection.
Measure: Number; unit: participants
Groups:
- Intervention Participants: Index participants in the intervention condition were trained to be Health Educators. The intervention focused on HIV risk reduction by teaching knowledge and skills to reduce injection, drug splitting, and sex risk, and by teaching communication skills to conduct outreach to personal risk network members. The intervention consisted of five group-based sessions, one individual session, and one dyad session with a risk network member.
- Control Participants: Index participants in the control condition attended groups that focused on injection drug-use related topics (e.g. HIV testing, Hepatitis C and drug overdose). The sessions were educational and did not include skills training. The control condition consisted of five group-based sessions.
Arm/Group | Intervention Participants | Control Participants
Number analyzed (Participants) | 101 | 95
participants | 2 | 21

5. Primary Outcome: Any Injection Risk (Monthly Versus Never)
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 70 | 76 | 191 | 138
participants | 15 | 27 | 79 | 53

6. Primary Outcome: Number of Needle or Cooker Sharers (2 or More Versus None)
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 82 | 82 | 212 | 280
participants | 5 | 17 | 37 | 31

7. Primary Outcome: Talked About HIV-related Topics With Drug Buddies (in the Past Month)
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 83 | 90 | 215 | 231
participants | 60 | 46 | 98 | 105

8. Primary Outcome: Showed a Needleless Syringe to Drug Buddies
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 94 | 100 | 244 | 302
participants | 78 | 16 | 35 | 55

9. Primary Outcome: Any Injection Risk (Monthly Versus Never)
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 81 | 83 | 227 | 166
participants | 12 | 25 | 63 | 46

10. Primary Outcome: Shared Cooker When Preparing Drugs
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 35 | 58 | 145 | 111
participants | 18 | 36 | 84 | 66

11. Primary Outcome: Number of Needle or Cooker Sharers (2 or More Versus None)
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 93 | 93 | 251 | 328
participants | 5 | 17 | 45 | 23

12. Primary Outcome: Injecting Drugs
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 99 | 107 | 281 | 354
participants | 35 | 58 | 143 | 108

13. Primary Outcome: Talked About HIV-related Topics With Drug Buddies (in Past Month)
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 68 | 84 | 219 | 265
participants | 44 | 35 | 96 | 106

14. Primary Outcome: Showed a Needleless Syringe to Drug Buddies
Time Frame: 18 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Number analyzed (Participants) | 100 | 107 | 286 | 360
participants | 84 | 22 | 37 | 67

15. Primary Outcome: Talked About Hepatitis to Drug Buddies
Time Frame: 18 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Intervention Participants | Control Participants
Number analyzed (Participants) | 95 | 100
participants | 51 | 29

ADVERSE EVENTS:
Arm/Group | Intervention Condition | Control Condition | Non-Randomized Baseline Index Participants | Risk Network Members
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/113 | 0/373 | 0/424
Other Adverse Events (participants affected / at risk) | 0/114 | 0/113 | 0/373 | 0/424

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No